CLINICAL TRIAL: NCT04260867
Title: Utility of Aromatherapy in Reducing Burnt Flesh Smell, Decreasing Intraoperative Anxiety, and Improving the Patient's Overall Experience During Cutaneous Surgical Procedures: a Randomized Controlled Trial
Brief Title: Essential Oils for Electrocautery
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Murad Alam, Professor of Dermatology, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STU00211721
Record Dates: First submitted 2020-02-06; First posted 2020-02-07 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — Oils, Volatile

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Aromatherapy (Experimental)
  Interventions: Other: Essential Oil
- Sham (Sham Comparator)
  Interventions: Other: No Essential Oil

INTERVENTIONS:
Other: Essential Oil — Those randomized to the treatment group will have containers filled with the essential oil of their choice.
  Arms: Aromatherapy
Other: No Essential Oil — Those randomized to the control group will then be given empty single-use handheld aromatherapy containers containing no essential oil.
  Arms: Sham

SUMMARY:
The purpose of this study is to assess whether essential oil aromatherapy could improve or eliminate the smell of burnt flesh from electrocautery and subsequently mitigate patient anxiety and discomfort during dermatologic skin surgery.

This is a randomized clinical trial. Approximately 210 electrocautery participants will be randomized to receive sham control/no aromatherapy or aromatherapy. Patients will be asked to complete a questionnaire after completion of the procedure to assess their experience. This study was a pilot study designed to determine the feasibility of this procedure.

Subjects currently living in the Chicago metropolitan area and meet inclusion/exclusion criteria will be invited and considered for enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. >18 years of age
2. Receiving same day cutaneous surgical procedure that requires electrocautery per protocol
3. In good general health as assessed by the investigator
4. Participants must have the ability to understand and the willingness to sign a written informed consent prior to registration on study

Exclusion Criteria:

1. Surgery site incompatible with the patient holding a handheld aromatherapy device (physician discretion)
2. Subject unwilling to sign an IRB approved consent form
3. Participants who are unable to communicate or cooperate with the investigator due to language problems, poor mental development, or impaired cerebral function are not eligible

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2020-12-22 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Self-reported perceptions of cautery smell on a 4-point likert scale | Immediately after surgery
  This is a patient-reported questionnaire about perceptions of smell.
Patient reported anxiety State-Trait Anxiety Inventory (STAI-6) | Immediately after surgery
  Patient perioperative anxiety will be reported on the 6-item shortform of the State-Trait Anxiety Inventory (STAI-6) directly after procedure

CONTACTS AND LOCATIONS:
Overall Officials: Murad Alam, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Department of Dermatology, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No